CLINICAL TRIAL: NCT01781702
Title: A Randomized, Double-blind, Multicenter, Phase 3 Study of Pelubiprofen Tab. & Celebrex Cap. for Comparative Evaluation of Safety & Efficacy in Rheumatoid Arthritis Patients
Brief Title: Phase 3 Study of Pelubiprofen Tab. & Celebrex Cap. in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: DW Plb RA301
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Pelubiprofen; Celebrex; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — pelubiprofen; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelubiprofen 30 mg (Experimental): Pelubiprofen 30 mg, tid
  Interventions: Drug: Pelubiprofen 30 mg
- Celebrex 200 mg (Active Comparator): Celebrex 200 mg, tid
  Interventions: Drug: Celebrex 200 mg

INTERVENTIONS:
Drug: Pelubiprofen 30 mg
  Arms: Pelubiprofen 30 mg
Drug: Celebrex 200 mg
  Arms: Celebrex 200 mg

SUMMARY:
A Randomized, Double-blind, Multicenter, Phase 3 Study of Pelubiprofen Tab. & Celebrex Cap. for Comparative Evaluation of Safety & Efficacy in Rheumatoid Arthritis Patients

ELIGIBILITY:
Inclusion Criteria:

1. Adult males/Females aged 18~80 years
2. Patient who are taking NSAIDs for the treatment of rheumatoid arthritis
3. Patients who belong to ACR functional class 1, 2, 3

Exclusion Criteria:

1. Patients who belong to ACR functional class 4
2. Patients who are hypersensitive to clinical trial medicines or excipient
3. Patients who have experience of Cerebrovascular bleeding, bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Changes in '100 mm pain VAS' value from baseline | -14, 0, 14, 28, 42 day

REFERENCES:
- [Derived] Choi IA, Baek HJ, Cho CS, Lee YA, Chung WT, Park YE, Lee YJ, Park YB, Lee J, Lee SS, Yoo WH, Song JS, Kang SW, Kim HA, Song YW. Comparison of the efficacy and safety profiles of a pelubiprofen versus celecoxib in patients with rheumatoid arthritis: a 6-week, multicenter, randomized, double-blind, phase III, non-inferiority clinical trial. BMC Musculoskelet Disord. 2014 Nov 18;15:375. doi: 10.1186/1471-2474-15-375. PMID 25403311